CLINICAL TRIAL: NCT00657631
Title: Acceptance and Commitment Therapy for Delusions
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Yulia Landa, Psy.D. Assistant Professor of Clinical Psychology, Weill Cornell Medical College
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0801009613
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2009-10

CONDITIONS: Schizophrenia; Delusional Disorder
Keywords: Acceptance and Commitment Therapy; Delusions
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Paranoid; Delusions | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Acceptance and Commitment Therapy will be administered to all subjects.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Considered part of the "third wave of CBT" along with Dialectical Behavior Therapy (DBT; Linehan, 1993) and Mindfulness-based Cognitive Therapy (MBCT; Segal, Williams, & Teasdale, 2001), ACT is built upon the strong, research-based foundation of CBT. However, while CBT for psychosis focuses on reducing symptoms, ACT focuses on changing the way in which the person experiences his or her symptoms so that the person can still live his or her life in accordance with his or her life values. Specifically, CBT attempts to reduce delusions by disputing the evidence for the delusion and ACT attempts to increase the person's ability to live his or her life while still experiencing delusions (Hayes, Strosahl & Wilson, 1999).
  Other Names: ACT

SUMMARY:
Symptoms of schizophrenia have historically been treatment resistant despite advances in psychopharmacology. Acceptance and Commitment Therapy (ACT) has been shown through some preliminary research to be effective with psychotic symptoms (Bach & Hayes, 2002). ACT is considered part of the "third wave of CBT" along with Dialectical Behavior Therapy (DBT; Linehan, 1993) and Mindfulness-based Cognitive Therapy (MBCT; Segal, Williams, & Teasdale, 2001). The target of change in ACT is acceptance of symptoms as experiences that a person can have without experiencing distress, and while living a life in accordance with one's values.

The current study assessed the effectiveness of ACT (8 sessions) for delusions. Participants received treatment as usual throughout the study. The intervention followed the protocol of ACT described in Hayes, Strosahl and Wilson (1999) in which treatment will consist of building acceptance, willingness, and commitment to change, clarifying values, defusion of thoughts and feelings, as well as defusion of self. These therapeutic aims attempted to be achieved by the practice of various exercises in and out of session as well as the discussion of various metaphors within session. It was hypothesized that participants will exhibit decreased distress due to delusions, decreased delusional conviction and a reduction of overall anxiety levels from participants' baselines.

DETAILED DESCRIPTION:
Four patients were recruited from New York Presbyterian Hospital, Weill Medical College, Payne Whitney Clinic (Manhattan Campus), outpatient psychiatric program. Patients were randomly assigned to a length of baseline before beginning the 8-week ACT treatment. There was be a five-week baseline period for all patients after which two patients will be introduced to ACT treatment in weekly increments. All patients received treatment as usual throughout baseline and ACT treatment. During baseline, patients were assessed by an independent rater every week and during ACT treatment, patients were assessed every other week and at a one-month follow-up. Each participant's assessment results were compared over time, so that there will be an established baseline level of functioning which will be compared to his or her level of functioning during treatment, at the end of treatment, and finally at the one-month follow-up. Hypotheses: It was hypothesized that patients' distress, anxiety and tension due to delusional thinking would decrease over time when comparing baseline to treatment, treatment to outcome, and then outcome to follow-up. Additionally, the number of delusional thoughts and the rate of re-hospitalization was hypothesized to decrease over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be considered for inclusion in the study if they meet DSM IV diagnostic criteria for:

  * Schizophrenia
  * Schizoaffective disorder
  * Schizophreniform Disorder
  * Delusional Disorder
  * Brief Psychotic Disorder
  * Psychotic Disorder NOS with current delusions (assessed via chart review)

Exclusion Criteria:

* Exclusion criteria include a current diagnosis of Mental Retardation
* Organic psychosis
* An inability to participant due to an acute medical condition
* Substance abuse within the past month, a high level of disorganization
* An inability to speak English
* Lack the ability to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
This study will illustrate how patients' distress due to delusional thinking decreases over time when comparing baseline to treatment, treatment to outcome, and then outcome to follow-up. | 4-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Landa, Psy.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College Oupatient Treatment Program of New York Presbyterian Hospital, New York, New York, United States

REFERENCES:
- [Background] Bach P, Hayes SC. The use of acceptance and commitment therapy to prevent the rehospitalization of psychotic patients: a randomized controlled trial. J Consult Clin Psychol. 2002 Oct;70(5):1129-39. doi: 10.1037//0022-006x.70.5.1129. PMID 12362963
- [Background] Linehan, M. M. (1993). Cognitive-behavioral treatment of borderline personality disorder. New York: Guilford Press.
- [Background] Segal, Z. V., Williams, J. M. G., & Teasdale, J. T. (2001). Mindfulness-based cognitive therapy for depression: A new approach to preventing relapse. New York: Guilford Press.
- [Background] Beck, A. T. (1976). Cognitive Therapy and the Emotional Disorders. New York: International Universities Press.
- [Background] Hayes, S. C., Strosahl, K. D. & Wilson, K. G. (1999). Acceptance and Commitment Therapy: An experiential approach to behavior change. New York: The Guilford Press.